CLINICAL TRIAL: NCT05947786
Title: Mpox Paediatric and Adolescent Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PENTA Foundation (Network)
Collaborators: University College, London (Other); European University Cyprus (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: VERDI MPOX paediatric study
Record Dates: First submitted 2023-05-26; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Monkey Pox; Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this multicentre, observational study on mpox in infants, children and adolescents is to increase knowledge about mpox infection and its associated disease in infants, children and adolescents. This will be done through the development of a harmonized system that will allow standard collection of information on demographics, clinical symptoms, clinical course, treatments and outcomes. The study will be carried out in three potential phases: Phase 1 entails the rapid development of an online paediatric registry collecting anonymised data from routine care on infants, children and adolescents with laboratory-confirmed mpox virus infection. If warranted, the study will proceed to Phase 2, an enhanced observational study of children and adolescents with confirmed mpox virus infection, if more detailed prospective data collection would aid the public health response. There is also the potential to initiate Phase 3, comprising of nested sub-studies to investigate specific research questions in this population.

DETAILED DESCRIPTION:
The primary objective of this multicentre observational study is to use a harmonised data system for the standard data collection and analysis to describe the presentation, clinical course and outcomes of laboratory-confirmed mpox virus infection in infants, children and adolescents by:

1. monitoring the temporal and geographical distribution of mpox infection in the paediatric and adolescent population, including in specific paediatric/adolescent groups, such as those with underlying conditions or with congenital mpox;
2. describing the epidemiology and clinical presentation of the disease, including outcomes of treatment administered as part of routine care;
3. describing high risk populations , including identifying factors associated with severe disease and death.

Phase 1 consists of the rapid development of an online registry for standard collection of data on infants, children and adolescents with laboratory-confirmed mpox infection, including adolescent girls who acquired mpox in pregnancy, and infants who acquired mpox through vertical transmission. All data will be fully anonymised, allowing rapid implementation in many countries without the need for ethics approval, where applicable.

If additional data collection would aid the public health response, the investigators might additionally include a second phase (Phase 2) of the project, with the aim to implement an enhanced prospective observational study of children and adolescents with confirmed mpox infection. This part of the project, if activated, will be a consented study collecting detailed data over the course of the disease.

Phase 3: initiation of nested sub-studies within the consented observational study (Phase 2) to investigate specific research questions in this population, including collection of samples, where necessary, for analysis and/or storage in a biobank. Each sub-study will require its own protocol and informed consent.

The database, networks and systems developed within Phases 1 to 3 will be flexible and designed to be readily adapted to data collection for other emerging and re-emerging infections in children.

ELIGIBILITY:
Inclusion Criteria:

* all infants, children and adolescents aged <18 years at the time of mpox diagnosis, with laboratory-confirmed mpox infection, as per national guidelines;
* mothers of eligible infants who are diagnosed with mpox at 28days or less are included in the study to collect maternal data on pregnancy and delivery

Exclusion Criteria:

* adolescents aged over 18 years old at mpox diagnosis.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants, children and adolescents with laboratory-confirmed mpox infection, including adolescent girls who acquired mpox in pregnancy, and infants who acquired mpox through vertical transmission.
  Phase 1 participants' consent may not be necessary as data collected is anonymous, phase 2 observational study participation would require participants'/ parent or legal representative consent as data collected is pseudonymised.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with severe mpox. | Throughout study completion, expected 2 years from study start.
  Severe mpox infection as measured by, for example, mortality, ICU admission, receipt of interventions

SECONDARY OUTCOMES:
Number of infants born to women infected with mpox in pregnancy, who are vertically infected with mpox. | Throughout study completion, expected 2 years from study start.
  Amongst infants born to women infected with mpox during pregnancy, the number who are themselves diagnosed with mpox within 28 days of birth.

CONTACTS AND LOCATIONS:
Locations (6):
- P. and A. Kyriakou Children's Hospital, Athens, Greece
- Spain (5):
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Niño Jesús, Madrid

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT05947786/Prot_000.pdf